CLINICAL TRIAL: NCT00961428
Title: Behavioral Assessment of the Reinforcing Effects of Exercise in Patients With Anorexia Nervosa
Brief Title: Motivation to Exercise in People With Anorexia Nervosa
Status: Completed | Type: Observational
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: #5544; K23MH071285-02 (NIH); NIMH K23 071285 (Other Grant/Funding Number: NIMH); DATR AK-TNAI1
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia Nervosa; Eating Disorders; Exercise; Physical Activity
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders; Motor Activity

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — fasting blood draws to measure cortison and leptin levels
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this research study is to determine the importance and level of physical activity in people with Anorexia Nervosa.

DETAILED DESCRIPTION:
A laboratory paradigm that uses a progressive ratio computerized work task will be used to determine the reinforcing value of exercise in hospitalized patients with AN, both before and after weight gain. In addition, we will examine the relationship between the reinforcing value of exercise and free-living physical activity in this population. We will also examine the relationship between the reinforcing value of exercise and measures of depression, anxiety, and cortisol, which we have found in previous studies to be associated with other measures of physical activity and exercise motivation. In order to determine whether physical activity in women with AN differs from that of non-eating disordered women, we will extend studies of physical activity to free-living control participants. All adult patients and controls will undergo body composition assessment once to measure the association between physical activity and percent body fat. Finally, to determine the impact of exercise reinforcement and physical activity on outcome in women with AN, we will conduct follow-up assessments in all patient participants for one year after discharge from the inpatient treatment unit."

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of Anorexia Nervosa (except amenorrhea)
* Female
* Age 18-45
* Medically Stable for exercise participation
* At a minimum of 75% Ideal Body Weight

Exclusion Criteria:

* Significant or current past medical illness including diabetes mellitis and heart disease
* Current or lifetime history or schizophrenia, bipolar disorder, or other psychotic disorder as defined by DSM-IV-TR
* Current suicidal ideation or recent suicidal behavior (within past 3 months)
* Drug or alcohol abuse in last 6 months
* Taking psychotropic medication
* Pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be patients with anorexia nervosa on the inpatient unit at New York State Psychiatric Institute
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
physical activity | Physical activity before and after weight restoration

CONTACTS AND LOCATIONS:
Overall Officials: B. Timothy Walsh, MD, Study Director — NYSPI; Evelyn Attia, MD, Principal Investigator — NYSPI
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States